CLINICAL TRIAL: NCT03222024
Title: Clinical Features, Management and Outcomes of Severe Ischaemic Stroke in Tertiary Hospitals in China: a Multi-centre Prospective Observational Study
Brief Title: Cohort Study for Severe Ischaemic Stroke
Acronym: SIS
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: Sichuan Academy of Medical Sciences (Other); The Affiliated Hospital Of Southwest Medical University (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); Chengdu University of Traditional Chinese Medicine (Other); Mianyang Central Hospital (Other); People's Hospital of Deyang City (Unknown); The First People's Hospital of Ziyang (Unknown); Jiangyou People's Hospital (Unknown); Science and Technology Department of Sichuan Province (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Simiao Wu, M.D., Ph.D., Dr, West China Hospital
Other Study IDs: 2017SZ0007
Record Dates: First submitted 2017-07-11; First posted 2017-07-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Severe Ischaemic Stroke; Malignant Ischaemic Stroke
Keywords: ischaemic stroke; severe; malignant; courses; risk factors; clinical course; management; prognosis
MeSH Terms: conditions — Ischemic Stroke; Lymphoma, Follicular; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — We will collect blood samples from patients with their written consent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe ischaemic stroke: patients with severe stroke on admission
  Interventions: Other: routine medical care
- Malignant ischaemic stroke: patients without severe stroke on admission but developing it in hospital
  Interventions: Other: routine medical care
- Mild to moderate ischaemic stroke: patients without severe stroke from onset to discharge
  Interventions: Other: routine medical care

INTERVENTIONS:
Other: routine medical care — This is an observational study for clinical course and outcomes of severe ischaemic stroke; therefore, interventions are prescribed by responsible doctors based on patients' clinical conditions, which is not interfered by current study

SUMMARY:
This is a multi-centre, prospective cohort study. The aim of this study is to investigate causes, risk factors, clinical course, management and outcomes of severe ischaemic stroke in a real-world setting in tertiary hospitals in China. Patients with acute ischaemic stroke from nine tertiary hospitals in western China will be recruited. Participants will be visited within 24 hours after admission, on day 3, day 7 and at discharge, to collect their clinical data, blood biomarkers, and brain imaging. A structured telephone interview will be conducted for each participant at 3 months and 1 year after stroke onset, respectively, to collect their functional outcomes. In-hospital outcomes include haemorrhagic transformation, brain oedema and death, 3-month and 1-year outcomes include survival status (death or survival) and functional outcome (scores of modified Rankin scale, mRS).

DETAILED DESCRIPTION:
Nine tertiary hospitals in Western China are participating in the study. In each participating hospital, stroke patients admitted to the Department of Neurology will be screened by their responsible doctors for eligibility. For patients who are potentially eligible, the doctor will introduce this study in detail with written information to the patient or their legal proxies. After participants (or their proxies) sign the consent form, investigators will collect their baseline data within 24 hours after admission (visit 1). Subsequent visits will be conducted on day 3 of admission or if the patient experiences neurological deterioration between visit 1 and day 3 (visit 2), on day 7 of admission or if neurological deterioration occurs between visit 2 and day 7 (visit 3), and on the day before discharge or on day 30 of admission, whichever is earlier (visit 4). At visit 1 investigators will record demographics, medical history, characteristics of current stroke, and results of the blood tests, brain imaging and other examinations, if applicable. At visit 4, investigators will record interventions and rehabilitation used during hospitalisation. At day 90 and 1 year of stroke onset, a trained investigator (neurologist) blind to all medical information will contact the participant to deliver a structured telephone interview and collect their functional outcomes.

Objectives of this study are: a) to explore causes of clinical worsening in acute ischaemic stroke, and for each type of clinical worsening to dynamically evaluate its clinical course and explore its risk factors; b) to explore the application of conventional stroke therapies in patients with severe ischaemic stroke in China; c) to investigate factors precipitating and predisposing malignant brain oedema following acute ischaemic stroke; and d) to better select patients with malignant brain oedema for individualised treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* Symptoms and signs of clinically definite acute stroke
* Time of stroke onset is known and within 30 days of admission
* CT or MRI brain scanning has reliably excluded both intracranial haemorrhage and structural brain lesions which can mimic stroke (e.g. brain tumour)

Exclusion Criteria:

* Likely to be unavailable for follow-up, e.g. no fixed home address
* Refuse to give consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischaemic stroke admitted to the Department of Neurology of nine participating hospitals will be included if they meet all inclusion criteria and do not have any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Functional outcome at 3 months after stroke onset | 3 months after stroke onset
  Modified Rankin scale score of patients at 3 months after the onset of ischaemic stroke.

SECONDARY OUTCOMES:
Proportion of patients with initially severe ischaemic stroke | 24 hours after admission
  Initially severe ischaemic stroke is defined as a) severe neurological deficits, assessed by the National Institute of Health Stroke Scale (NIHSS) scored 15 or over, b) loss of consciousness, assessed by the Glasgow Coma Scale (GCS) scored 8 or less, or item 1a of NIHSS scored 1 or over, or c) intubation, mechanical ventilation, or admitted to intensive care unit on admission.
Proportion of patients experiencing clinical worsening following acute ischaemic stroke | 30 days after admission
  Clinical worsening is defined as a) neurological deterioration with an increase of NIHSS score of 4 or more as compared to baseline NIHSS, b) a decline of consciousness, which leads to a GCS score of 8 or less, or item 1a of NIHSS scored 1 or over, c) need for invasive interventions such as hemicraniectomy, or d) death in hospital.
Proportion of patients with malignant brain oedema following acute ischaemic stroke | 30 days after admission
  Malignant brain oedema is defined as symptoms or signs of clinical worsening associated with imaging evidence of space-occupying brain oedema.
Clinical course of stroke severity in patients with initially severe stroke | 30 days after admission
  Dynamically record scores of National Institute of Health Stroke Scale (NIHSS) from day 0, day 3, day 7 to day 30 after admission.
Changes in consicousness level of patients with initially severe stroke from day 0, day 3, day 7 to day 30 after admission. | 30 days after admission
  Dynamically record scores of Glasgow Coma Scale (GCS)
Functional outcome at 1 year after stroke onset | 1 year after stroke onset
  Modified Rankin scale score of patients at 1 year after the onset of ischaemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Liu, MD, Study Chair — West China Hospital; Shihong Zhang, MD, Study Director — West China Hospital; Simiao Wu, MD, PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu S, Yuan R, Xiong Y, Zhang S, Wu B, Liu M. Clinical features, management and outcomes of severe ischaemic stroke in tertiary hospitals in China: protocol for a prospective multicentre registry-based observational study. BMJ Open. 2018 Oct 28;8(10):e024900. doi: 10.1136/bmjopen-2018-024900. PMID 30373783
- [Background] Wu S, Yuan R, Wang Y, Wei C, Zhang S, Yang X, Wu B, Liu M. Early Prediction of Malignant Brain Edema After Ischemic Stroke. Stroke. 2018 Dec;49(12):2918-2927. doi: 10.1161/STROKEAHA.118.022001. PMID 30571414
- [Derived] Wu S, Wang Y, Yuan R, Liu M, Hua X, Huang L, Guo F, Yang D, Li Z, Wu B, Wang C, Duan J, Ling T, Zhang H, Zhang S, Wu B, Zhu C, Anderson CS, Liu M. Clinical course, causes of worsening, and outcomes of severe ischemic stroke: A prospective multicenter cohort study. Chin Med J (Engl). 2025 Jul 5;138(13):1578-1586. doi: 10.1097/CM9.0000000000003556. Epub 2025 Mar 17. PMID 40090964
- [Derived] Wu S, Wang Y, Yuan R, Guo F, Yang D, Li Z, Wu B, Wang C, Duan J, Ling T, Zhang H, Zhang S, Wu B, Anderson CS, Liu M. Predicting the emergence of malignant brain oedema in acute ischaemic stroke: a prospective multicentre study with development and validation of predictive modelling. EClinicalMedicine. 2023 Apr 27;59:101977. doi: 10.1016/j.eclinm.2023.101977. eCollection 2023 May. PMID 37152361